CLINICAL TRIAL: NCT03405064
Title: A Phase III, Multi-centre, Randomized Study to Compare the Efficacy and Safety of Levonadifloxacin (IV and Oral) With Linezolid (IV and Oral) in Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Brief Title: Comparative Study of Levonadifloxacin (IV and Oral) With Linezolid (IV and Oral) in Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W-771/2349-301
Record Dates: First submitted 2017-11-22; First posted 2018-01-19 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Acute Bacterial Skin and Skin Structure Infections
MeSH Terms: interventions — levonadifloxacin; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- levonadifloxacin (Experimental): oral levonadifloxacin (1000 mg BID) or IV levonadifloxacin (800 mg BID)
  Interventions: Drug: Oral Levonadifloxacin/Linezolid Tablet; Drug: Intravenous Levonadifloxacin/Linezolid Infusion
- linezolid (Active Comparator): oral linezolid (600 mg BID) or IV linezolid (600 mg BID)
  Interventions: Drug: Oral Levonadifloxacin/Linezolid Tablet; Drug: Intravenous Levonadifloxacin/Linezolid Infusion

INTERVENTIONS:
Drug: Oral Levonadifloxacin/Linezolid Tablet — oral levonadifloxacin (1000 mg BID) or oral linezolid (600 mg BID)
Drug: Intravenous Levonadifloxacin/Linezolid Infusion — IV levonadifloxacin (800 mg BID) or IV linezolid (600 mg BID)

SUMMARY:
This is a phase III, multi-center, randomized, active-comparator, study in subjects with ABSSSI. The study has two subgroups for assessment of efficacy and safety - oral subgroup 1 and IV subgroup 2. Each subgroup will comprise of two treatment arms.

DETAILED DESCRIPTION:
Subjects willing to participate in the study and fulfilling all eligibility criteria will receive either oral therapy (subgroup 1) or IV therapy (subgroup 2). The investigator can initiate treatment with either oral or IV therapy based on clinical judgement i.e subjects who require IV therapy (like subjects with severe ABSSSI or where oral administration is not feasible).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to participate in the study and provide a written informed consent
* Subjects with ABSSSI characterized by any of the following infection types:

  1. Cellulitis/erysipelas: diffuse skin infection characterized by spreading areas of redness, edema, and/or induration
  2. Wound infection: An infection characterized by purulent drainage from a wound with surrounding redness, edema, and/or induration
  3. Major cutaneous abscess: An infection characterized by a collection of pus within the dermis or deeper that is accompanied by redness, edema, and/or induration
* Subjects with lesion size area of at-least 75 cm2. Lesion size will be measured by the area of redness, edema, or induration
* Subjects with suspected and/or documented evidence of Gram-positive infection

Exclusion Criteria:

* 1. ABSSSI meeting any of the following criteria:

  1. Severely impaired arterial blood supply (such that the likelihood of amputation of the infected anatomical site is likely)
  2. ABSSSI expected to require more than 10 days of antimicrobial therapy as per the discretion of the Investigator
  3. Subject with suspected or confirmed osteomyelitis or septic arthritis or gangrene
  4. ABSSSI requiring surgical intervention (except surgical incision and drainage for abscess) 2. Subjects who have received prior antibiotic therapy within past 24 hours for the treatment of current episode of ABSSSI. Following are the exceptions to this criteria:

  <!-- -->

  1. Subjects who received a single dose of a short-acting antibacterial drug within 24 hours of enrolment
  2. Subjects with evidence of clinical progression of ABSSSI while on antibacterial drug therapy after at-least 48 hours
  3. Subjects who received an antibacterial drug for surgical prophylaxis and subsequently develop ABSSSI 3. Subjects with current history or diagnosis of HIV, positive test result for hepatitis B surface antigen (HBsAg) or Hepatitis C virus (HCV) 4. Subjects with any clinically significant abnormalities in pulmonary, gastrointestinal, endocrine, hepatic or renal systems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
The non-inferiority of oral levonadifloxacin with oral linezolid in ABSSSI by measuring the Overall Clinical Response at Test of Cure (TOC) visit in modified Intentto-treat (mITT) population in oral treatment subgroups | 0-14 days
To establish the non-inferiority of IV levonadifloxacin with IV linezolid in ABSSSI measuring the Overall Clinical Response at Test of Cure (TOC) visit in modified Intentto-treat (mITT) population in IV treatment subgroups | 0-14 days

SECONDARY OUTCOMES:
The safety of oral and IV levonadifloxacin based on adverse events reported, vital signs and physical examination findings, clinical laboratory evaluation, and ECG collected during the study. | 0-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Chugh, MD, Study Director — Wockhardt
Locations (32):
- India (32):
  - Osmania General Hospital, Hyderabad, Andhra Pradesh
  - Government General Hospital (Associated by Government Siddhartha Medical College), Vijayawada, Andhra Pradesh
  - Sanjivani Superspeciality Hospital Pvt. Ltd., Ahmedabad, Gujarat
  - Medistar Multispeciality Hospital Pvt.Ltd., Himmatnagar, Gujarat
  - GMERS Medical College & General Hospital, Vadodara, Gujarat
  - Parul Institute of Medical Science, Vadodara, Gujarat
  - Victoria Hospital, Bangalore, Karnataka
  - Vinaya Hospital and Research Centre, Mangalore, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - Government Medical College, Kozhikode, Kerala
  - Ishwar Institute of Healthcare, Aurangabad, Maharashtra
  - TNMC & BYL Nair Hospital, Mumbai, Maharashtra
  - LTM Medical College and General Hospital, Mumbai, Maharashtra
  - Government Medical College and Hospital, Nagpur, Maharashtra
  - Shree Hospital & Critical Care Centre, Nagpur, Maharashtra
  - Rahate Surgical Hospital, Nagpur, Maharashtra
  - Cresent Hospital and Heart Centre, Nagpur, Maharashtra
  - Indira Gandhi Government Medical College and Hospital, Nagpur, Maharashtra
  - B.J. Medical College and Sassoon General Hospital, Pune, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Oyster & Pearl Hospital, Pune, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Lifepoint Hospital, Pune, Maharashtra
  - Datta Meghe Institute of Medical Sciences (Deemed University) Jawaharlal Nehru Medical College, Wardha, Maharashtra
  - S.R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - SMS Hospital, Jaipur, Rajasthan
  - Marudhar Hospital, Jaipur, Rajasthan
  - M.V. Hospital & Research Centre, Lucknow, Uttar Pradesh
  - Ajanta Research Centre, Lucknow, Uttar Pradesh
  - KRM Hospital and Research Centre, Lucknow, Uttar Pradesh
  - Popular Hospital, Varanasi, Uttar Pradesh
  - Om Surgical & Maternity Home, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatia A, Mastim M, Shah M, Gutte R, Joshi P, Kumbhar D, Periasamy H, Palwe SR, Chavan R, Bhagwat S, Patel M, Llorens L, Friedland HD. Efficacy and Safety of a Novel Broad-Spectrum Anti-MRSA Agent Levonadifloxacin Compared with Linezolid for Acute Bacterial Skin and Skin Structure Infections: A Phase 3, Openlabel, Randomized Study. J Assoc Physicians India. 2020 Aug;68(8):30-36. PMID 32738837